CLINICAL TRIAL: NCT06907225
Title: Physiological Responses to Heat Stress During High-risk Events
Status: Enrolling by invitation | Type: Observational
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gabrielle Giersch, Research Physiologist, United States Army Research Institute of Environmental Medicine
Other Study IDs: 24-29
Record Dates: First submitted 2025-03-24; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-01

CONDITIONS: Thermoregulation
Keywords: Thermoregulation; Heat illness
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood and urine samples (without DNA) will be retained for biological analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: None-placebo — None - observational study

SUMMARY:
Exertional heat stroke (EHS) affects ~500 Military Personnel and over 100 Soldiers every year, and it is believed that these numbers are underreported. EHS is the most severe form of exertional heat illness (EHI) and can result in substantial, long-lasting organ damage, and even death in severe cases. Based on current knowledge and training needs, it is impossible to prevent every EHS - which shifts the focus from exclusively prevention to a combination of prevention, treatment, and enhancing recovery as much as possible. While many risk factors have been identified and there are adequate treatments available, biomarkers associated with heat stroke risk, recovery, and return-to-duty (RTD) remain largely unclear. The purpose of the proposed study is to enhance knowledge surrounding biomarkers of EHS and long-term health consequences that result from EHS. The investigators will recruit research volunteers for a field study in order to collect pre-, post-, and follow-up measures from a high-risk EHS event (i.e. ruck marches, timed runs) this will allow us to have a basis for comparison between Soldiers who collapse with EHS (from previously collected data) and those that complete high-risk events, but do not collapse. This will allow for comparison between the groups to identify EHS-specific biomarkers that could aid in recovery and RTD decisions for Soldiers.

DETAILED DESCRIPTION:
Exertional heat stroke (EHS) affects ~500 Military Personnel (MSMR, 2022) and over 100 Soldiers (Giersch et al, 2022) every year. EHS is the most severe form of exertional heat illness and can result in substantial, long-lasting organ damage and sometimes death. While some risk factors for EHS are known (Roberts et al, 2021), and the investigators have effective treatments available (Caldwell et al, 2022), EHS cases are not 100% preventable. Furthermore, it is not possible to investigate EHS directly in the laboratory, as safety criteria limit the core temperatures (Tcore) permitted. Therefore, clinicians must rely on prospective clinical investigations after normal training or events (e.g. road races, marathons, etc.).

Collecting data on Soldiers who experience heat stroke helps further our understanding of potential predisposing factors, recovery, and long-term health consequences. Specifically, biomarkers of cardiac, kidney, muscle, and liver damage can inform recovery and return-to-duty (RTD) decisions, but the direct effect of EHS on these systems remains largely unknown. Recent discussions with international colleagues, including the Surgeon General of the Israeli Defense Force, highlight the need for a prospective identification of those at greatest risk for EHS (BG Elon Glassberg, Surgeon General, Israeli Defense Force, personal communication, September 2022).

The proposed study will utilize a similar approach as that employed by a previous study (Kenney et al, 2012), that examined serum creatine kinase (CK) levels in a cohort of healthy basic trainees at Fort Moore. While 200 IU/L is commonly the upper limit of normal values, they found that trainees often had CK values exceeding 1,000 IU/L, which reflects chronic high-intensity physical training, rather than a pathological condition such as exertional rhabdomyolysis (ER). The findings from this paper have influenced the diagnostic criteria for ER, such that a CK level of 50x the upper limit of normal is often required for diagnosis. The effect, if any, of chronic/routine high intensity physical training on other biomarkers, such as creatinine for acute kidney injury and alanine aminotransferase/aspartate aminotransferase (ALT/AST) for liver injury, is unknown. Knowledge of the 'normal' physiological response to exercise-heat stress, as assessed by biomarkers of end-organ function, may potentially guide healthcare providers diagnostic decision-making process and prevent over-diagnosis of conditions. This in turn may result in shorter limited duty time and improved readiness. The proposed investigation will utilize a similar approach, but in a cohort relevant to EHS.

Whereas most EHS cases occur during ruck marches and timed runs (DeGroot et al, MSMR 2022), what is less clear is what represents a "positive" or adaptive physiological response to these high-risk events. One of the goals of the present project will be to identify biomarkers of "successful" exposure to high-risk events. These biomarkers would be present in individuals who successfully complete the events, but don't experience an exertional heat illness (effectively acting as a healthy control to EHS cases). The prospective quantification of differences between EHS cases and healthy controls could provide insights into useful biomarkers (including markers of kidney, liver, and cardiac injury) to differentiate between patients and aid in the identification and treatment of EHS. The results of this study, therefore, will likely contribute to the identification of EHS-specific biomarkers or biomarker levels (i.e. clinical values) to develop better guidance for prevention, treatment and return-to-duty.

If successful, this work can be followed up by investigating treatments for EHS and their response to biomarkers immediately following hyperthermia and during recovery. Identifying the recovery period for these biomarkers in healthy individuals following high risk events will yield greater knowledge in EHS specific biomarkers and recovery. Follow-on work could also investigate EHS severity and the spectrum of exertional heat injuries to evaluate risk and prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (to include cis- and transgender males and females and nonbinary) 18 years of age or greater
* Current military service (active, Reserve, or National Guard)
* Currently participating in training

Exclusion Criteria:

* Females who are pregnant
* Any individual currently on a physical profile that restricts running or foot marching
* History of obstructive disease of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis.
* Scheduled MRI within 2 weeks after core temp pill ingestion
* Known allergies to skin adhesive
* Blood donation in the past 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample population included in this investigation will be that of Soldiers undergoing high-risk training events in military training. There are no gender, race, or ethnicity limitations.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Core temperature | Collected only during training, pre-exercisce, post-exercise, and after recovery (from 0-36 hours)
  Body temperature recorded during training
Creatinine from blood serum | Measured at least once every 6 hours for up to 36 hours
  Serum creatinine measures to evaluate kidney function
Alanine aminotransferase from blood samples | Measured at least once every 6 hours for up to 36 hours
  Measure of liver function (ALT) from blood
Aspartate aminotransferase (AST) | Measured at least once every 6 hours for up to 36 hours
  Liver function measure (AST) from blood
Heart rate | Measured during training only from start of training up to completion (~4 hours)
  Heart rate measured during activity

SECONDARY OUTCOMES:
Urinary KIM-1 | Measured at least once every 6 hours for up to 36 hours
  Measure of kidney function (KIM-1) from urine
Urinary creatinine | Measured at least once every 6 hours for up to 36 hours
  Kidney function measures (creatinine) from urine
Blood sodium concentration | Measured at least once every 6 hours for up to 36 hours
  Blood sodium concentration

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fort Novosel, Fort Novosel, Alabama
  - Field Study, Fort Jackson, South Carolina

IPD SHARING:
Plan to Share IPD: No
Not permitted to share as Army data

REFERENCES:
- [Background] Roberts WO, Armstrong LE, Sawka MN, Yeargin SW, Heled Y, O'Connor FG. ACSM Expert Consensus Statement on Exertional Heat Illness: Recognition, Management, and Return to Activity. Curr Sports Med Rep. 2021 Sep 1;20(9):470-484. doi: 10.1249/JSR.0000000000000878. PMID 34524191
- [Background] Williams VF, Oh GT. Update: Heat illness, active component, U.S. Armed Forces, 2021. MSMR. 2022 Apr 1;29(4):8-14. PMID 35608520